CLINICAL TRIAL: NCT00198588
Title: Open-Label Trial to Evaluate the Efficacy and Safety of the Use of Argatroban in Patients With Heparin-Induced Thrombocytopenia
Brief Title: Efficacy and Safety Study of Argatroban to Treat Heparin-Induced Thrombocytopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Haruko Yamamoto, National Cardiovascular Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARG-HIT-CVD
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Heparin-Induced Thrombocytopenia
Keywords: heparin-induced thrombocytopenia; argatroban; cardiac surgery; acute coronary syndrome; thrombosis; amputation; anticoagulation
MeSH Terms: conditions — Acute Coronary Syndrome; Thrombosis | interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: argatroban — beginning dose: 0.7microgram/kg/H

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of argatroban in the patients with heparin-induced thrombocytopenia (HIT)/ HIT and thrombosis syndrome (HITTS). This multi-center trial covers mainly the patients with cardiovascular diseases. Subjects are included in the trial when they are clinically diagnosed of HIT/HITTS. Initial dose of argatroban is 0.7μg/kg/min, which is about one-third of the approved dose in the US. The reason of the lower initial dose is that the approved dose of argatroban in Japan (for the treatment of ischemic stroke) is about 0.7μg/kg/min and safety of higher doses of the drug are not confirmed. A sub-study of pharmacokinetics is simultaneously conducted to reveal the relationship among the dose, aPTT, and blood drug concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Males of non-pregnant females >=20 and <=80 years of age
2. Those with the diagnosis of HIT or HITTS made by the following diagnostic criteria, or those who have positive results of HIT antibody

   * diagnostic criteria of HIT
   * a fall in platelet count to less than 100,000/μL or a 50% decrease in platelets after the initiation of heparin therapy with no apparent explanation other than HIT
   * diagnostic criteria of HITTS

     * those who met the diagnosis criteria of HIT
     * presence of an arterial or venous thrombosis documented by appropriate imaging technique (ultrasound, angiography etc.) or supported by clinical evidence such as a myocardial infarction, stroke, pulmonary embolism, or other clinical indications of vascular occlusion(absence of pulse, cold, cyanotic extremities, etc.)
   * patients with history of HIT/HITTS with positive test results (HIT antibody or platelet function test) could be enrolled without present thrombocytopenia
3. patients willing and able to give informed consent

Exclusion Criteria:

1. any condition which in the investigator's opinion, contraindicated the use of argatroban or endangered the patient if he or she participated in this trial
2. clinically significant or uncontrolled endocrine, renal, pulmonary, gastrointestinal, or psychiatric disorder of sufficient severity that the investigator deemed antithrombotic therapy with argatroban to be contraindicated
3. unexplained aPTT>200% of control at baseline
4. documented coagulation disorder or unexplained bleeding diathesis unrelated to HIT
5. lumbar puncture within the past 7 days
6. known clinical site of bleeding. Patients with a known site of clinical bleeding could be enrolled if the investigator deemed the risk of continued thrombosis outweighed the potential bleeding risk
7. serious liver disfunction
8. females of known or suspected pregnancy
9. breast feeding females
10. participation in other clinical drug trials within the past 30 days
11. history of hypersensitivity to argatroban
12. concomitant use of cimetidine
13. previous participation in this trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-06; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Death, new thrombosis, amputation | till 37 days

SECONDARY OUTCOMES:
Achievement of anticoagulation therapy | till 37 days
Improvement of thrombocytopenia | till 37 days

CONTACTS AND LOCATIONS:
Overall Officials: Hitonobu TOMOIKE, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (20):
- Japan (20):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Hakodate National Hospital, Hakodate, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kurume University Hospital, Kurume, Hukuoka
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City General Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Kyoto Second Red Cross Hospital, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - National Cardiovascular Center, Suita, Osaka
  - Sakakibara Memorial Hospital, Fuchū, Tokyo
  - The University of Tokyo Hospital, Tokyo, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo, Tokyo
  - Keio University Hospital, Tokyo, Tokyo
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni, Yamaguchi
  - Yamaguchi University Hospital, Ube, Yamaguchi